CLINICAL TRIAL: NCT05817799
Title: Impact of Hemodialysis on Plasma Carnitine Levels in Patients With End Stage Renal Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bahria University (Other)
Collaborators: Pakistan Navy Station Shifa Hospital (Other); Jinnah Postgraduate Medical Centre (Other Government); University of Karachi (Other)
Responsible Party: Principal Investigator, Sadia Rehman, Senior Assistant Professor, Bahria University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ERC 2022/23
Record Dates: First submitted 2023-03-24; First posted 2023-04-18 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Hemodialysis Complication
Keywords: Hemodialysis; L-Carnitine; chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Carnitine

STUDY DESIGN:
Intervention Model Description: Subjects of group B oral intervention group were given oral L-carnitine supplementation in the form of L-Carnitine tablets 500 mg thrice daily under strict monitoring for 5 months. The vitals were monitored daily during the course of supplementation.
  Subjects of group B intravenous group were given Intra venous L-Carnitine as a dose of 20mg/kg IV bolus infused over 2-3 minutes, administered into intra venous line after every hemodialysis session ( thrice a week) for 5 months.
  Complete general physical examination was done on every dialysis session. Patients were strictly monitored for the development of any signs of distress during the course of supplementation the drug. The patients and their attendants were educated about monitoring the vitals at home daily and to inform nephrologist immediately in case of any signs of allergy or distress. The supplementation was given after obtaining ethical approval and informed consent and under direct supervision of a Nephrologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental): L-Carnitine 500mg thrice daily
  1g L-Carnitine IV three times a week
  Interventions: Drug: L-Carnitine 500Mg thrice daily; Drug: 1g L-Carnitine IV three times a week
- control (No Intervention): no intervention given

INTERVENTIONS:
Drug: L-Carnitine 500Mg thrice daily — L-Carnitine 500mg oral thrice daily
  Arms: intervention
Drug: 1g L-Carnitine IV three times a week — 1g IV L-Carnitine three times a week
  Arms: intervention

SUMMARY:
OBJECTIVES

* To assess the levels of plasma carnitine in controls and hemodialysis patients.
* To give supplementary L-carnitine to study subjects for a duration of 5months.
* To compare the values of plasma carnitine before and after L carnitine supplementation.
* To assess the role of carnitine supplementation on biochemical and clinical parameters.

DETAILED DESCRIPTION:
.ABSTRACT INTRODUCTION Dialysis therapy can cause a decrease in both free carnitine and plasma acyl carnitines after only six months of dialysis treatment. A positive correlation between AC/FC ratio and months on HD therapy has been reported. We investigate in this study the role of oral L-carnitine supplementation on anemia, blood pressure, cardiac dysfunction and muscle cramps in hemodialysis patients.

OBJECTIVES

* To assess the levels of plasma carnitine in controls and hemodialysis patients.
* To give supplementary L-carnitine to study subjects for a duration of 5months.
* To compare the values of plasma carnitine before and after L carnitine supplementation.
* To assess the role of carnitine supplementation on biochemical and clinical parameters.

STUDY DESIGN AND SETTING: It will be a case-control study, which will be conducted in the Department of Biochemistry, University of Karachi in collaboration with Nephrology ward of JPMC, Karachi in a period of one year after approval of synopsis.

METHOD: Total 120 subjects will be included in this study which will be divided into two groups. Group A will comprise of 60 subjects of Chronic renal failure who will be the control group. Group B will comprise of 60 subjects who will be on hemodialysis for more than 1 year. Blood samples will be taken after informed consent. Group B subjects will be given L-Carnitine supplementation for five months under strict monitoring. Physical, biochemical and clinical parameters of group B subjects will be compared before and after supplementation.

RESULTS: Data will be analyzed using SPSS version 21. Results will be shared after completion of research.

CONCLUSION: conclusion will be shared after completion of research.

ELIGIBILITY:
Inclusion Criteria: • Individuals of either sex (male and female).

* The study included people between the ages of 18 and 50 who had had dialysis for more than two years without taking additional antioxidants.

Exclusion Criteria:

* • Individuals with any other chronic ailment, such as cancer or tuberculosis.

  * Patients with acute renal failure who are receiving hemodialysis.
  * All subjects who refused to take part in the investigation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-02 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
L-Carnitine levels in hemodialysis | 5 months
  plasma carnitine will be detected before and after giving intervention (unit μmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Sadia Rehman, Principal Investigator — Bahria University Health Sciences, Karachi
Locations (1):
- Jinnah Post Graduate Medical Center, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Hurot JM, Cucherat M, Haugh M, Fouque D. Effects of L-carnitine supplementation in maintenance hemodialysis patients: a systematic review. J Am Soc Nephrol. 2002 Mar;13(3):708-714. doi: 10.1681/ASN.V133708. PMID 11856775
- [Result] Kuwasawa-Iwasaki M, Io H, Muto M, Ichikawa S, Wakabayashi K, Kanda R, Nakata J, Nohara N, Tomino Y, Suzuki Y. Effects of L-Carnitine Supplementation in Patients Receiving Hemodialysis or Peritoneal Dialysis. Nutrients. 2020 Nov 1;12(11):3371. doi: 10.3390/nu12113371. PMID 33139659
- [Result] Zhu Y, Xue C, Ou J, Xie Z, Deng J. Effect of L-carnitine supplementation on renal anemia in patients on hemodialysis: a meta-analysis. Int Urol Nephrol. 2021 Oct;53(10):2149-2158. doi: 10.1007/s11255-021-02835-5. Epub 2021 Mar 13. PMID 33713287
- [Result] Maruyama T, Maruyama N, Higuchi T, Nagura C, Takashima H, Kitai M, Utsunomiya K, Tei R, Furukawa T, Yamazaki T, Okawa E, Ando H, Kikuchi F, Abe M. Efficacy of L-carnitine supplementation for improving lean body mass and physical function in patients on hemodialysis: a randomized controlled trial. Eur J Clin Nutr. 2019 Feb;73(2):293-301. doi: 10.1038/s41430-018-0348-y. Epub 2018 Oct 23. PMID 30353121
- [Result] Huang H, Song L, Zhang H, Zhang H, Zhang J, Zhao W. Influence of L-carnitine supplementation on serum lipid profile in hemodialysis patients: a systematic review and meta-analysis. Kidney Blood Press Res. 2013;38(1):31-41. doi: 10.1159/000355751. Epub 2014 Feb 6. PMID 24525835
- [Result] Hamedi-Kalajahi F, Imani H, Mojtahedi S, Shabbidar S. Effect of L-Carnitine Supplementation on Inflammatory Markers and Serum Glucose in Hemodialysis Children: A Randomized, Placebo-Controlled Clinical Trial. J Ren Nutr. 2022 Mar;32(2):144-151. doi: 10.1053/j.jrn.2021.03.009. Epub 2021 Nov 3. PMID 34740538
- [Derived] Rehman S, Farhan M, Kumar S, Sarfraz MR, Naveed A, Khan MT, Huq H. Efficacy of Intravenous Versus Oral Administration of Levocarnitine in Maintenance Hemodialysis Patients: A Randomized Controlled Trial Investigating Therapeutic Approaches to Renal Anemia. Health Sci Rep. 2025 Jan 5;8(1):e70297. doi: 10.1002/hsr2.70297. eCollection 2025 Jan. PMID 39763581